CLINICAL TRIAL: NCT03328364
Title: A Registry Based Study Evaluating Overall Survival and Treatment Length in mCRPC Patients Treated With Enzalutamide in Sweden
Status: Completed | Type: Observational
Sponsor: Astellas Pharma a/s (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9785-MA-3166
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: enzalutamide; metastatic castration-resistant prostate cancer; Xtandi; registry based study; MDV3100; mCRPC
MeSH Terms: interventions — enzalutamide; Docetaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- enzalutamide (mCRPC pre-chemo): Patients treated with enzalutamide prior to chemotherapy
  Interventions: Drug: enzalutamide
- enzalutamide and chemotherapy (mCRPC post chemo): Patients treated with enzalutamide who have previously undergone treatment with chemotherapy (docetaxel)
  Interventions: Drug: enzalutamide; Drug: docetaxel

INTERVENTIONS:
Drug: enzalutamide — oral
  Other Names: Xtandi; MDV3100
Drug: docetaxel — intravenous infusion
  Groups: enzalutamide and chemotherapy (mCRPC post chemo)

SUMMARY:
The purpose of this study is to provide real world data on treatment with enzalutamide in metastatic castration-resistant prostate cancer (mCRPC) patients.

The primary purpose is to evaluate overall survival (OS) in mCRPC patients treated with enzalutamide who have previously undergone treatment with chemotherapy (docetaxel) (post chemo patients).

This study will also evaluate treatment duration with enzalutamide in patients pre- and post-chemo.

DETAILED DESCRIPTION:
The data source in this study is a local hospital registry created from a patient follow up of prostate cancer patients.

ELIGIBILITY:
Inclusion criteria:

* Chemo naïve mCRPC patients treated with enzalutamide and ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration).
* mCRPC patients treated with enzalutamide and ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration) post chemo.

Exclusion Criteria

* mCRPC patients previously exposed to Radium-223, abiraterone acetate and/or cabazitaxel for mCRPC (pre- and post chemotherapy).
* Patients previously exposed to chemotherapy or abiraterone acetate+prednisolone in combination with GnRH analogue for hormone sensitive prostate cancer (HSPC).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mCRPC initiating treatment with enzalutamide pre- and post- chemo registered in the prostate cancer registry.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-24 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Overall survival in metastatic castration-resistant prostate cancer (mCRPC) patients treated with enzalutamide, who have previously undergone treatment with chemotherapy (docetaxel) | Up to a maximum of four years
  Overall survival is defined as time from initiation to death of any cause.

SECONDARY OUTCOMES:
Treatment duration of enzalutamide in pre chemo mCRPC patients | Up to a maximum of four years
  Treatment duration is defined as time from initiation to treatment discontinuation of any cause.
Treatment duration of enzalutamide in post chemo mCRPC patients | Up to a maximum of four years
  Treatment duration is defined as time from initiation to treatment discontinuation of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Scientific Advisor, Study Chair — Astellas Pharma a/s
Locations (1):
- Site SE46001, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Alghazali M, Lofgren A, Jorgensen L, Svensson M, Fagerlund K, Bjartell A. A registry-based study evaluating overall survival and treatment duration in Swedish patients with metastatic castration-resistant prostate cancer treated with enzalutamide. Scand J Urol. 2019 Oct;53(5):312-318. doi: 10.1080/21681805.2019.1657494. Epub 2019 Sep 6. PMID 31815592
- See also: Link to results on ACSR web site — https://astellasclinicalstudyresults.com/study.aspx?ID=337